CLINICAL TRIAL: NCT01126970
Title: A Double-Blind, Multi-Center, Randomized, Parallel-Group Study to Assess the Efficacy and Safety of 400 mg of Velneperit (S-2367) and 120 mg of Orlistat Administered Individually or Combined Orally Three Times Per Day With a Reduced Calorie Diet (RCD) in Obese Subjects
Brief Title: Double-Blind, Multi-Center, Randomized Study to Assess the Efficacy and Safety of Velneperit (S-2367) and Orlistat Administered Individually or Combined With a Reduced Calorie Diet (RCD) in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002A2828
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: reduced calorie diet; orlistat; velneperit
MeSH Terms: conditions — Obesity | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebos. (Placebo Comparator): Velneperit Placebo q.d.+ Orlistat Placebo t.i.d.
  Interventions: Drug: Orlistat Placebo; Drug: Velneperit Placebo; Other: Reduced Calorie Diet
- Velneperit 400 mg (Experimental): Velneperit 400 mg q.d.
  Interventions: Drug: Velneperit 400 mg; Drug: Orlistat Placebo; Other: Reduced Calorie Diet
- Orlistat 120 mg (Active Comparator): Orlistat 120 mg t.i.d.
  Interventions: Drug: Orlistat 120 mg; Drug: Velneperit Placebo; Other: Reduced Calorie Diet
- Velneperit 400 mg + Orlistat 120 mg (Experimental): Velneperit 400 mg q.d.and Orlistat 120 mg t.i.d
  Interventions: Drug: Velneperit 400 mg; Drug: Orlistat 120 mg; Other: Reduced Calorie Diet

INTERVENTIONS:
Drug: Velneperit 400 mg — Velneperit 400 mg q.d.
  Other Names: S-2367
  Arms: Velneperit 400 mg; Velneperit 400 mg + Orlistat 120 mg
Drug: Orlistat 120 mg — Orlistat 120 mg t.i.d
  Other Names: Xenical
  Arms: Orlistat 120 mg; Velneperit 400 mg + Orlistat 120 mg
Drug: Orlistat Placebo — Orlistat Placebo t.i.d.
  Arms: Placebos.; Velneperit 400 mg
Drug: Velneperit Placebo — Velneperit Placebo q.d
  Arms: Orlistat 120 mg; Placebos.
Other: Reduced Calorie Diet — Reduced calorie diet

SUMMARY:
To evaluate the weight loss effect and safety of 400 mg velneperit and 120 mg orlistat administered individually or combined three times per day for 24 weeks while on a reduced calorie diet (RCD) and also to evaluate the steady-state trough concentrations of velneperit (S-2367), velneperit (S-2367) tert-butyl OH, and velneperit (S-2367) tert-butyl OH-O glucuronide following 400 mg of velneperit (S-2367) three times per day and 120 mg of orlistat, either combined or separate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age at the time of informed consent
* Body mass index (BMI) of 30.0 to 45.0 kg/m2 inclusive. BMI for study inclusion must be obtained from the Interactive Voice Response System/Web Response System (IVRS/WRS). (Visit 1 body weight and height obtained prior to the single-blind period will be used by the IVRS/WRS in the calculation.)
* Weight that has not fluctuated by more than 3% for the 90 days prior to Visit 1
* Non-smoker and no use of tobacco or nicotine products for at least 1 year prior to Visit 1
* Normotensive or acceptable level of hypertension, defined as systolic <160 and diastolic <95 mmHg
* No clinically significant laboratory abnormalities
* Negative urine drug screen for drugs of abuse
* No clinically significant findings on medical history, physical examination, and electrocardiogram (ECG) and no known history of clinically significant ECG abnormalities
* Negative serum pregnancy test in women of child-bearing potential (Females must be at least one year post-partum.)
* Males either should remain abstinent, be sterile or agree to use an approved method of contraception (which for males includes use of a condom with spermicide) Visit 1 through 12 weeks following the last dose, in addition to having a female partner use an effective form of contraception as noted below
* All female subjects must be non-pregnant (confirmed by a negative serum pregnancy test), have no plans of becoming pregnant during the study, and must be at least one year post-partum, non-lactating, postmenopausal, (defined as cessation of regular menstrual periods for at least one year and confirmed by a follicle-stimulating hormone test), or surgically sterile by hysterectomy and/or bilateral oophorectomy or tubal ligation. Females of child-bearing potential must agree to use acceptable forms of birth control including oral, implantable or transdermal contraceptives; or use of one of the following double-barrier methods: intrauterine device with spermicide, diaphragm with spermicide, cervical cap with spermicide, female condom with spermicide, or a male condom with spermicide by the male sexual partner
* Able to comply with all required study procedures and schedule
* Able to speak and read English
* Signed and dated informed consent form prior to any study-related procedures

Exclusion Criteria:

* Obesity of known endocrine or genetic origin (eg, hypothyroidism, Cushing's syndrome or diagnosed polycystic ovarian syndrome) meeting one of the following conditions:

  * Menstrual irregularity due to oligo- or anovulation
  * Evidence of hyperandrogenism, whether clinical (hirsutism, acne, or male pattern balding) or biochemical (high serum androgen concentrations)
  * Exclusion of other causes of hyperandrogenism and menstrual irregularity, such as congenital adrenal hyperplasia, androgen-secreting tumors, and hyperprolactinemia]
* History of malignancy within the previous 5 years with the exception of non-melanoma skin cancer or surgically cured cervical cancer
* Human immunodeficiency virus (HIV) identified by history or previous HIV test
* Any serious medical condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study including any clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs
* Known history or evidence of a psychiatric disorder that in the opinion of the investigator would preclude the subject from participating in the trial. Stable or controlled anxiety or depression are permitted. Treatment with an antidepressant or anxiolytic drug is permitted if in accordance with Appendix 4. Subjects with a score of 11 or higher on the depression portion of the Hospital Anxiety and Depression Scale are excluded.
* Subjects with pancreatitis or chronic pancreatic inflammation
* History of Type 1 or Type 2 diabetes mellitus as defined by HbA1c > 6.5% or blood glucose values of > 126 mg/dl or treated Type 2 diabetes mellitus
* Any weight gain during the single-blind lead-in period (Visit 1 and Visit 3)
* History of surgical or device (eg, gastric bypass) intervention for obesity surgery, stomach banding surgery, or any other surgical procedure(s) that attempt to promote/aid weight loss. Note: Liposuction will be allowed if done more than 90 days prior to screening
* History of alcoholism or drug addiction/substance abuse within 1 year of Visit 1. Note: No alcohol consumption is permitted within 48 hours prior to blood collections for analysis of lipid profiles.
* Abnormal thyroid stimulating hormone level at screening
* Subjects with hypothyroidism
* Subjects with genetic hematologic disease or trait with or without manifestation of disease.
* Use of chronic medications/products within 90 days prior to Visit 1 or during the study that are known to cause weight gain. Investigators will discuss with the Sponsor's Medical Monitor any concomitant medications about which they are uncertain.
* Use of systemic corticosteroids or Depo Provera®
* History of fenfluramine or dexfenfluramine (Fen-Phen) administration (except with a prior documented echocardiogram showing no valvular abnormalities.)
* History of participation in any weight loss program within 90 days prior to Visit 1
* Participation in any weight loss medication/product study in which receipt of weight loss medication/product occurred within 90 days prior to Visit 1
* Use of any prescription or nonprescription over the counter medication/product or herbal/phytotherapeutic/plant-derived medications/products for weight loss, appetite suppression, weight control or treat obesity (includes investigational products) within 90 days prior to Visit 1 or during the study
* Subjects with cholestasis or chronic malabsorption
* Donation of blood or blood products 90 days prior to Visit 1 or during the study
* Exposure to an investigative medication within the past 30 days or 5 half-lives, whichever is longer or concurrent participation in any clinical trial
* Previous velneperit (S-2367) or other neuropeptide Y (NPY) Y5 agonist or antagonist use
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study
* Positive Hepatitis B or C serology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the change from baseline in body weight (kg) over the 168-day (24-week) double-blind treatment period, where baseline body weight was defined as the last measurement prior to randomization | 168 days (24 weeks)
  Change in body weight from baseline to 24 weeks

SECONDARY OUTCOMES:
Efficacy analysis: The proportion of subjects with (a) a 5% decrease in body weight at Visit 7 and Visit 10 and (b) percent change in body weight from baseline to each study visit was summarized by treatment group | change from baseline to each study visit
  Percentage of subjects who achieve a 5% decrease in body weight
Efficacy analysis: The change in waist & hip circumference (cm) from baseline to each study visit was summarized by treatment group | Change from baseline to each study visit
  Change in physical measurement from baseline
Efficacy analysis: The proportion of subjects with a decrease equal to or greater than 1 BMI unit at Visit 7 and Visit 10 was summarized by treatment group | Baseline to Visits 7 and 10
  The proportion of subjects with decreases in BMI of 1 unit
Safety analysis: (a) Treatment-emergent adverse events and (b) monitoring clinical laboratory evaluations, vital signs, 12-lead electrocardiograms, and physical examinations | Baseline to each visit and to Week 24
  Change from baseline to each visit and to Week 24

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Santa Rosa, California
  - Waterbury, Connecticut
  - Clearwater, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Ponte Vedra, Florida
  - Augusta, Georgia
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Milford, Massachusetts
  - North Dartmouth, Massachusetts
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Albuquerque, New Mexico
  - Manlius, New York
  - Rochester, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Greenville, South Carolina
  - Nashville, Tennessee
  - New Braunfels, Texas
  - Renton, Washington
  - Wauwatosa, Wisconsin